CLINICAL TRIAL: NCT00385736
Title: A Multicenter, Randomized, Double-blind Placebo-controlled Study of the Human Anti-TNF Monoclonal Antibody Adalimumab for the Induction of Clinical Remission in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Efficacy and Safety of Adalimumab in Subjects With Moderately to Severely Acute Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Roopal B Thakkar, M.D., Project Director, Global Pharmaceutical Research and Development, Humira Gastroenterology, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-826; 2006-002781-20 (EudraCT Number)
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Results first posted 2010-05-27 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Ulcerative Colitis
Keywords: Moderate to Severe Ulcerative Colitis; Double-blind; Adalimumab; Induction of Clinical Remission
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adalimumab 80/40 (Experimental)
  Interventions: Biological: adalimumab
- Adalimumab 160/80/40 (Experimental)
  Interventions: Biological: adalimumab
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: adalimumab — Prefilled syringe, 40 mg (loading dose then every other week dosing). 80 mg at Week 0, 40 mg at Week 2, and 40 mg every other week starting at Week 4.
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab 80/40
Biological: adalimumab — Prefilled syringe, 40 mg (loading dose then every other week dosing). 160 mg at Week 0, 80 mg at Week 2, and 40 mg every other week starting at Week 4.
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab 160/80/40
Biological: placebo — Placebo for 40 mg syringe. Matching placebo for loading dose and every other week dosing. Subjects received placebo at Weeks 0, 2, 4, and 6, followed by 160 mg adalimumab at Week 8, 80 mg adalimumab at Week 10, and 40 mg adalimumab eow thereafter (prior to Amendment 3) or 40 mg adalimumab eow starting at Week 8 (after Amendment 3).
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the efficacy and safety of adalimumab for the induction of clinical remission in subjects with moderately to severely active ulcerative colitis.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, randomized, double-blind (DB), placebo-controlled trial designed to evaluate the efficacy and safety of the human anti-TNF monoclonal antibody adalimumab for the induction of clinical remission in participants with moderately to severely active ulcerative colitis (UC).

Adult participants with moderate to severe UC (Mayo score of 6 to 12 points with endoscopy subscore of 2 to 3 points), confirmed by colonoscopy with biopsy or by flexible sigmoidoscopy with biopsy, were enrolled at 80 sites worldwide. The study enrolled 576 participants, including 186 participants under the original protocol and protocol Amendments 1 and 2, and 390 participants under protocol Amendments 3 and 4.

Participants enrolled in the study prior to Amendment 3 were randomized in a 1:1 ratio to receive adalimumab or placebo during the 12-week DB induction period. Participants received 4 injections of adalimumab 40 mg (160 mg) or 4 injections of placebo at Baseline (Week 0), followed by 2 injections of adalimumab 40 mg (80 mg) or 2 injections of placebo at Week 2, followed by 1 injection of adalimumab 40 mg or placebo at Weeks 4 and 6. At Week 8, participants randomized to placebo received 4 injections of adalimumab 40 mg (160 mg) followed by 2 injections of adalimumab 40 mg (80 mg) at Week 10. Participants randomized to adalimumab received 3 injections of placebo and 1 injection of adalimumab 40 mg at Week 8 and 1 injection of placebo and 1 injection of adalimumab 40 mg at Week 10. All participants continued to receive 1 injection of open-label (OL) adalimumab 40 mg every other week beginning at Week 12 up to Week 52 (or the early termination visit). Starting at Week 14, participants who had inadequate responses to treatment (as defined using partial Mayo scores) were permitted to dose escalate to adalimumab 40 mg weekly. Participants with persistent inadequate response while on weekly treatment could be discontinued from the study at the discretion of the investigator.

In August 2007, the study design was amended to incorporate an additional adalimumab induction dosing arm of 80/40 mg. Earlier that year, both 160/80-mg and 80/40-mg induction regimens had been approved in the EU as induction treatment for Crohn's disease. The adalimumab induction dosing regimen of 80/40 mg was therefore included so that both of these approved induction regimens would be evaluated for the induction of remission of UC.

Participants enrolled in the study after Amendment 3 were randomized in a 1:1:1 ratio to receive adalimumab (1 of 2 regimens) or placebo during the 8-week DB induction period. Participants received DB therapy from Baseline until Week 8 and OL therapy from Week 8 until the end of the study. In the first adalimumab dosing arm (adalimumab 80/40), participants received 2 injections of adalimumab 40 mg (80 mg) and 2 injections of placebo at Baseline followed by 1 injection of adalimumab 40 mg and 1 injection of placebo at Week 2, and 1 injection of adalimumab 40 mg every other week thereafter. In the second adalimumab DB induction dosing arm (adalimumab 160/80), participants received 4 injections of adalimumab 40 mg (160 mg) at Baseline followed by 2 injections of adalimumab 40 mg (80 mg) at Week 2, and 1 injection of adalimumab 40 mg every other week thereafter. Participants randomized to placebo received 4 injections of placebo at Baseline followed by 2 injections of placebo at Week 2, and 1 injection of placebo at Weeks 4 and 6. Beginning at Week 8, but after the Week 8 study assessments had been completed, all participants received 1 injection of OL adalimumab 40 mg every other week until Week 52 or early termination. Starting at Week 12, participants who had inadequate responses to treatment (as defined using partial Mayo scores) were permitted to dose escalate to adalimumab 40 mg weekly. Participants with persistent inadequate response while on weekly treatment could be discontinued from the study at the discretion of the investigator.

For the analysis of efficacy parameters during the DB Period through Week 8, only participants randomized under Protocol Amendment 3 or later were considered ("Efficacy Analysis Set - Induction" in the participant flow). For the analysis of efficacy parameters during the OL Period through Week 52, all randomized participants (under any version of the protocol) who received at least 1 dose of study drug were considered ("Efficacy Analysis Set - Maintenance" in the participant flow). For the analysis of safety parameters, all participants who received at least 1 dose of study drug were considered ("Safety Analysis Set" in the participant flow).

Twelve ranked secondary variables during the DB Period through Week 8 were to be tested in a hierarchical order to account for multiple testing. These variables are identified as "Ranked Secondary Endpoints" in the results section below. Additionally, non-ranked secondary variables during the OL Period through Week 52 were tested and are presented after the ranked secondary endpoints in the results section below.

ELIGIBILITY:
The following eligibility criteria applied to participants enrolled following Amendment 3 to the study protocol.

Inclusion Criteria:

1. Male and female participants >= 18 years of age
2. Diagnosis of ulcerative colitis for greater than 90 days prior to Baseline
3. Diagnosis of active ulcerative colitis confirmed by colonoscopy with biopsy or flexible sigmoidoscopy with biopsy during the Screening Period, with exclusion of infection
4. Active UC with a Mayo score of 6 to 12 points and endoscopy subscore of 2 to 3 points, despite concurrent treatment with at least 1 of the following (oral corticosteroids or immunosuppressants or both as defined below):

   * Stable oral corticosteroid dose (prednisone dose of >= 20 mg/day or equivalent) for at least 14 days prior to Baseline or stable oral corticosteroid dose (prednisone of < 20 mg/day) for at least 40 days prior to Baseline.

   and/or
   * At least a consecutive 90 day course of azathioprine or 6-mercaptopurine (6 MP) prior to Baseline, with a dose of azathioprine >= 1.5 mg/kg/day or 6 MP >= 1 mg/kg/day (rounded to the nearest available tablet formulation), or a dose that is the highest tolerated by the participant (e.g., due to leukopenia, elevated liver enzymes, nausea) during that time. Participant was to be on a stable dose for at least 28 days prior to Baseline.

   Concurrent therapy was not required for participants who were previously treated with corticosteroids or immunosuppressants (azathioprine or 6-MP) during the previous 5 years and, in the judgment of the investigator, have failed to respond to or could not tolerate their treatment.
5. Had to be able to self-administer or has caregiver who can reliably administer subcutaneous injections.
6. Had to be able and willing to give written informed consent and to comply with the requirements of this study protocol.
7. Female had to be either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or of childbearing potential and practicing an approved method of birth control throughout the study and for 150 days after last dose of study drug. Examples of approved methods of birth control included the following:

   * Condoms, sponge, foams, jellies, diaphragm or intrauterine device
   * Oral, parenteral or intravaginal contraceptives for 90 days prior to study drug administration
   * A vasectomized partner
8. The results of the serum pregnancy test performed at the Screening Visit and urine pregnancy test performed at the Baseline Visit had to be negative.
9. Judged to be in generally good health as determined by the principal investigator

Exclusion Criteria:

1. History of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, or ileostomy for ulcerative colitis or is planning bowel surgery.
2. Received infliximab or any other anti-TNF agent or any biological therapy in the past.
3. Received previous treatment with adalimumab or previous participation in an adalimumab clinical study.
4. Received cyclosporine, tacrolimus, or mycophenolate mofetil within 30 days prior to Baseline.
5. Received intravenous corticosteroids within 14 days prior to Screening or during the Screening Period.
6. Received therapeutic enema or suppository, other than required for endoscopy, within 14 days prior to the Screening endoscopy and during the remainder of the Screening Period.
7. Current diagnosis of fulminant colitis and/or toxic megacolon.
8. Participants with disease limited to the rectum (ulcerative proctitis).
9. Current diagnosis of indeterminate colitis.
10. Current diagnosis and/or history of Crohn's disease.
11. Currently receiving total parenteral nutrition.
12. Discontinued use of azathioprine or 6-MP within 28 days of Baseline.
13. Discontinued use of corticosteroid within 14 days of Baseline.
14. Participants using aminosalicylates for less than 90 days prior to Baseline, not on a stable dose for at least 28 days prior to Baseline, or discontinued use within 28 days of Baseline.
15. Participants with positive Clostridium difficile stool assay.
16. Infections requiring treatment with intravenous (IV) antibiotics, IV antivirals, or IV antifungals within 30 days prior to Baseline or oral antibiotics, oral antivirals, or oral antifungals within 14 days prior to Baseline.
17. History of malignancy other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix. If the Screening colonoscopy/flexible sigmoidoscopy showed evidence of dysplasia or a malignancy, the participant was not to be enrolled in the study.
18. History of listeria, histoplasmosis, chronic or active hepatitis B infection, human immunodeficiency virus, immunodeficiency syndrome, central nervous system demyelinating disease, or untreated tuberculosis (TB).
19. Female participants who was pregnant or breast-feeding or considering becoming pregnant during the study. There should be at least a 150-day period between the last dose of study drug and either conception or initiation of breast-feeding in women of childbearing potential.
20. Poorly controlled medical condition(s), such as uncontrolled diabetes, unstable ischemic heart disease, moderate to severe congestive heart failure, recent cerebrovascular accident and any other condition, which in the opinion of the investigator, would put the participant at risk by participation in the protocol.
21. Received any investigational agent within 30 days or 5 half lives prior to Baseline (whichever is longer).
22. History of clinically significant drug or alcohol abuse during the previous year.
23. Participants with known hypersensitivity to the excipients of adalimumab as stated in the label.
24. Participants with any prior exposure to Tysabri® (natalizumab).
25. Participants currently taking both budesonide and prednisone (or equivalent) simultaneously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2006-11; Primary Completion 2009-04 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Thakkar, MD, Study Director — Abbott
Locations (80):
- United States (29):
  - Site Ref # / Investigator 2080, Birmingham, Alabama
  - Site Ref # / Investigator 6034, Mobile, Alabama
  - Site Ref # / Investigator 5100, Fayetteville, Arkansas
  - Site Ref # / Investigator 5390, Orange, California
  - Site Ref # / Investigator 5392, San Diego, California
  - Site Ref # / Investigator 2245, Bridgeport, Connecticut
  - Site Ref # / Investigator 2240, Gainesville, Florida
  - Site Ref # / Investigator 2230, South Miami, Florida
  - Site Ref # / Investigator 5393, Atlanta, Georgia
  - Site Ref # / Investigator 2231, Atlanta, Georgia
  - Site Ref # / Investigator 2498, Chicago, Illinois
  - Site Ref # / Investigator 2078, Chevy Chase, Maryland
  - Site Ref # / Investigator 2238, Silver Springs, Maryland
  - Site Ref # / Investigator 1971, Boston, Massachusetts
  - Site Ref # / Investigator 2246, Rochester, Minnesota
  - Site Ref # / Investigator 2243, Kansas City, Missouri
  - Site Ref # / Investigator 2247, Mexico, Missouri
  - Site Ref # / Investigator 2233, Lincoln, Nebraska
  - Site Ref # / Investigator 2236, Cedar Knolls, New Jersey
  - Site Ref # / Investigator 2072, New York, New York
  - Site Ref # / Investigator 2241, Charlotte, North Carolina
  - Site Ref # / Investigator 2232, Raleigh, North Carolina
  - Site Ref # / Investigator 11801, Wilmington, North Carolina
  - Site Ref # / Investigator 2074, Cincinnati, Ohio
  - Site Ref # / Investigator 2126, Cleveland, Ohio
  - Site Ref # / Investigator 6090, Germantown, Tennessee
  - Site Ref # / Investigator 2076, Nashville, Tennessee
  - Site Ref # / Investigator 2229, Bellevue, Washington
  - Site Ref # / Investigator 2077, Milwaukee, Wisconsin
- Austria (7):
  - Site Ref # / Investigator 4936, Graz
  - Site Ref # / Investigator 6224, Hall in Tirol
  - Site Ref # / Investigator 3830, Innsbruck
  - Site Ref # / Investigator 7508, Linz
  - Site Ref # / Investigator 3829, Salzburg
  - Site Ref # / Investigator 4937, Vienna
  - Site Ref # / Investigator 3831, Vienna
- Belgium (3):
  - Site Ref # / Investigator 3861, Bonheiden
  - Site Ref # / Investigator 3859, Liège
  - Site Ref # / Investigator 3862, Roeselare
- Canada (5):
  - Site Ref # / Investigator 2224, Calgary, Alberta
  - Site Ref # / Investigator 2227, Edmonton, Alberta
  - Site Ref # / Investigator 2226, Vancouver, British Columbia
  - Site Ref # / Investigator 2223, Winnipeg, Manitoba
  - Site Ref # / Investigator 2138, Toronto, Ontario
- Czechia (5):
  - Site Ref # / Investigator 3858, Brno
  - Site Ref # / Investigator 3856, Olomouc
  - Site Ref # / Investigator 3857, Ostrava
  - Site Ref # / Investigator 3854, Prague
  - Site Ref # / Investigator 3855, Prague
- Germany (6):
  - Site Ref # / Investigator 3832, Berlin
  - Site Ref # / Investigator 13983, Essen
  - Site Ref # / Investigator 3834, Jena
  - Site Ref # / Investigator 3833, Kiel
  - Site Ref # / Investigator 3878, Mainz
  - Site Ref # / Investigator 3897, Munich
- Hungary (3):
  - Site Ref # / Investigator 3852, Budapest
  - Site Ref # / Investigator 3850, Budapest
  - Site Ref # / Investigator 3849, Győr
- Italy (5):
  - Site Ref # / Investigator 3876, Bologna
  - Site Ref # / Investigator 3848, Milan
  - Site Ref # / Investigator 3845, Palermo
  - Site Ref # / Investigator 6232, Rome
  - Site Ref # / Investigator 3846, Rome
- Netherlands (2):
  - Site Ref # / Investigator 3873, Eindhoven
  - Site Ref # / Investigator 3875, Leiden
- Poland (3):
  - Site Ref # / Investigator 8061, Lodz
  - Site Ref # / Investigator 13804, Sopot
  - Site Ref # / Investigator 8055, Warsaw
- Puerto Rico (2):
  - Site Ref # / Investigator 2392, Ponce
  - Site Ref # / Investigator 2393, San Juan
- Slovakia (7):
  - Site Ref # / Investigator 3839, Banská Bystrica
  - Site Ref # / Investigator 3838, Bratislava
  - Site Ref # / Investigator 3841, Bratislava
  - Site Ref # / Investigator 3842, Nitra
  - Site Ref # / Investigator 14721, Prešov
  - Site Ref # / Investigator 14521, Trenčín
  - Site Ref # / Investigator 3840, Trnava
- Sweden (3):
  - Site Ref # / Investigator 8503, Gothenburg
  - Site Ref # / Investigator 8504, Linköping
  - Site Ref # / Investigator 8502, Lund

REFERENCES:
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- [Derived] Feagan BG, Sandborn WJ, Lazar A, Thakkar RB, Huang B, Reilly N, Chen N, Yang M, Skup M, Mulani P, Chao J. Adalimumab therapy is associated with reduced risk of hospitalization in patients with ulcerative colitis. Gastroenterology. 2014 Jan;146(1):110-118.e3. doi: 10.1053/j.gastro.2013.09.032. Epub 2013 Sep 22. PMID 24067881
- [Derived] Reinisch W, Sandborn WJ, Panaccione R, Huang B, Pollack PF, Lazar A, Thakkar RB. 52-week efficacy of adalimumab in patients with moderately to severely active ulcerative colitis who failed corticosteroids and/or immunosuppressants. Inflamm Bowel Dis. 2013 Jul;19(8):1700-9. doi: 10.1097/MIB.0b013e318281f2b7. PMID 23665965
- [Derived] Reinisch W, Sandborn WJ, Hommes DW, D'Haens G, Hanauer S, Schreiber S, Panaccione R, Fedorak RN, Tighe MB, Huang B, Kampman W, Lazar A, Thakkar R. Adalimumab for induction of clinical remission in moderately to severely active ulcerative colitis: results of a randomised controlled trial. Gut. 2011 Jun;60(6):780-7. doi: 10.1136/gut.2010.221127. Epub 2011 Jan 5. PMID 21209123

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Treatment group received placebo at Weeks 0, 2, 4, and 6, followed by 160 mg adalimumab at Week 8, 80 mg adalimumab at Week 10, and 40 mg adalimumab thereafter (prior to Amendment 3) or 40 mg adalimumab eow starting at Week 8 (after Amendment 3).
- Adalimumab 80/40: Treatment group received 80 mg at Week 0, 40 mg at Week 2, and 40 mg every other week starting at Week 4.
- Adalimumab 160/80/40: Treatment group received 160 mg at Week 0, 80 mg at Week 2, and 40 mg every other week starting at Week 4.
Period: Efficacy Analysis Set - Induction
Arm/Group | Placebo | Adalimumab 80/40 | Adalimumab 160/80/40
Started | 130 (Enrolled under Amendment 3 or 4 of the protocol.) | 130 (Enrolled under Amendment 3 or 4 of the protocol.) | 130 (Enrolled under Amendment 3 or 4 of the protocol.)
Completed | 121 (Completed Week 8 of the study.) | 118 (Completed Week 8 of the study.) | 121 (Completed Week 8 of the study.)
Not Completed | 9 | 12 | 9
Not completed — Adverse Event | 5 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Lack of Efficacy | 4 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Other | 0 | 0 | 1
Period: Efficacy Analysis Set - Maintenance
Arm/Group | Placebo | Adalimumab 80/40 | Adalimumab 160/80/40
Started | 222 (Includes all subjects with confirmed UC enrolled since the start of the study) | 130 (Includes all subjects with confirmed UC enrolled since the start of the study) | 223 (Includes all subjects with confirmed UC enrolled since the start of the study)
Completed | 153 | 86 | 143
Not Completed | 69 | 44 | 80
Not completed — Adverse Event | 23 | 15 | 23
Not completed — Withdrawal by Subject | 6 | 6 | 14
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Lack of Efficacy | 38 | 16 | 31
Not completed — Protocol Violation | 2 | 1 | 6
Not completed — Other | 0 | 4 | 4
Period: Safety Analysis Set
Arm/Group | Placebo | Adalimumab 80/40 | Adalimumab 160/80/40
Started | 223 (Includes all subjects enrolled since the start of the study.) | 130 (Includes all subjects enrolled since the start of the study.) | 223 (Includes all subjects enrolled since the start of the study.)
Completed | 153 | 86 | 143
Not Completed | 70 | 44 | 80
Not completed — Adverse Event | 23 | 15 | 23
Not completed — Withdrawal by Subject | 6 | 6 | 14
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Lack of Efficacy | 38 | 16 | 31
Not completed — Protocol Violation | 2 | 1 | 6
Not completed — Other | 1 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab 80/40 | Adalimumab 160/80/40 | Total
Number analyzed (Participants) | 130 | 130 | 130 | 390
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 1 | 4
  Between 18 and 65 years | 125 | 120 | 124 | 369
  >=65 years | 4 | 8 | 5 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 38.9 (12.68) | 41.6 (13.99) | 38.2 (13.46) | 39.5 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 47 | 147
  Male | 82 | 78 | 83 | 243
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 41 | 103
  Slovakia | 12 | 22 | 13 | 47
  Austria | 7 | 11 | 5 | 23
  Italy | 11 | 6 | 7 | 24
  Czech Republic | 23 | 11 | 18 | 52
  Hungary | 9 | 3 | 7 | 19
  Canada | 26 | 25 | 20 | 71
  Belgium | 4 | 2 | 2 | 8
  Poland | 2 | 2 | 2 | 6
  Germany | 3 | 14 | 9 | 26
  Netherlands | 1 | 4 | 0 | 5
  Sweden | 0 | 0 | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Clinical Remission Per Mayo Score at Week 8
Description: Clinical remission per Mayo score is defined as a total Mayo score <= 2 and no individual subscore > 1.
  The Mayo Score is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 12 (severe disease) and is a composite of 4 subscores:
  Stool Frequency Subscore, Rectal Bleeding Subscore, Endoscopy Subscore, and Physician's Global Assessment Subscore, each of which ranges from 0 (normal) to 3 (severe disease).
Time Frame: Week 8
Population: All participants enrolled after Amendment 3 to the study protocol (which introduced the adalimumab 80/40 treatment arm) and who received at least 1 dose of study drug were included in this intent-to-treat (ITT) analysis. Nonresponder imputation (NRI) was used.
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 80/40 | Adalimumab 160/80/40
Number analyzed (Participants) | 130 | 130 | 130
Proportion of participants | 9.2 | 10.0 | 18.5
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 160/80/40; Test type: Superiority or Other; p = 0.031, Chi-squared — The primary endpoint analysis was carried out in hierarchical order (as presented) to handle the multiplicity issues induced by the two adalimumab groups being compared to placebo and to control the overall alpha level of 0.05
Statistical Analysis 2: Comparison: Placebo vs Adalimumab 80/40; Test type: Superiority or Other; p = 0.833, Chi-squared — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Ranked Secondary Endpoint #1: Proportion of Participants With Clinical Response Per Mayo Score at Week 8 (Adalimumab 160/80/40 Versus Placebo).
Description: Clinical response per Mayo score is defined as a decrease in Mayo score of >= 3 points and >= 30% from Baseline, plus either a decrease in rectal bleeding subscore of >= 1 point or an absolute rectal bleeding subscore of 0 or 1.
  The Mayo Score is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 12 (severe disease) and is a composite of 4 subscores:
  Stool Frequency Subscore, Rectal Bleeding Subscore, Endoscopy Subscore, and Physician's Global Assessment Subscore, each of which ranges from 0 (normal) to 3 (severe disease).
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 160/80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 44.6 | 54.6
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 160/80/40; Test type: Superiority or Other; p = 0.107, Chi-squared — Ranked secondary analyses were carried out in hierarchical order (as presented) to handle the multiplicity issues and to control the overall alpha level of 0.05

3. Secondary Outcome: Ranked Secondary Endpoint #2: Proportion of Participants With Mucosal Healing at Week 8 (Adalimumab 160/80/40 Versus Placebo).
Description: Mucosal healing is defined as Endoscopy Subscore of 0 or 1 as assessed by flexible sigmoidoscopy. Possible scores range from 0-3 as follows:
  0 = Normal or inactive disease, 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 2 = Moderate disease (marked erythema, absent vascular pattern, friability, erosions), 3 = Severe disease (spontaneous bleeding, ulceration)
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 160/80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 41.5 | 46.9
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 160/80/40; Test type: Superiority or Other; p = 0.382, Chi-squared — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Ranked Secondary Endpoint #3: Proportion of Participants With Rectal Bleeding Subscore Indicative of Mild Disease (<= 1) at Week 8 (Adalimumab 160/80/40 Versus Placebo).
Description: Rectal Bleeding Subscore ranges from 0-3 as follows:
  0 = no blood seen, 1 = streaks of blood with stool less than half the time, 2 = obvious blood with stool most of the time, 3 = blood alone passed
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 160/80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 66.2 | 77.7
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 160/80/40; Test type: Superiority or Other; p = 0.038, Chi-squared — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Ranked Secondary Endpoint #4: Proportion of Participants With Physician's Global Assessment Subscore Indicative of Mild Disease (<= 1) at Week 8 (Adalimumab 160/80/40 Versus Placebo).
Description: The Physician's Global Assessment Subscore acknowledges the 3 other subscores (Stool Frequency, Rectal Bleeding, and Endoscopy), the subject's daily record of abdominal discomfort and functional assessment, and other observations such as physical findings and the subject's performance status. Possible scores range from 0-3 as follows:
  0 = Normal (other subscores are 0), 1 = Mild disease (other subscores are mostly 1), 2 = Moderate disease (other subscores are 1 to 2), 3 = Severe disease (other subscores are 2 to 3)
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 160/80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 46.9 | 60.0
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 160/80/40; Test type: Superiority or Other; p = 0.035, Chi-squared — [p-value comment as in outcome 2, analysis 1]

6. Secondary Outcome: Ranked Secondary Endpoint #5: Proportion of Participants With Stool Frequency Subscore Indicative of Mild Disease (<= 1) at Week 8 (Adalimumab 160/80/40 Versus Placebo).
Description: Stool Frequency Subscore ranges from 0-3 as follows: 0 = Normal number of stools for this participant, 1 = 1-2 stools more than normal, 2 = 3-4 stools more than normal, 3 = 5 or more stools more than normal
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 160/80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 37.7 | 48.5
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 160/80/40; Test type: Superiority or Other; p = 0.080, Chi-squared — [p-value comment as in outcome 2, analysis 1]

7. Secondary Outcome: Ranked Secondary Endpoint #6: Proportion of Participants With Clinical Response Per Mayo Score at Week 8 (Adalimumab 80/40 Versus Placebo).
Description: as for outcome 2
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 44.6 | 51.5
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80/40; Test type: Superiority or Other; p = 0.264, Chi-squared — [p-value comment as in outcome 2, analysis 1]

8. Secondary Outcome: Ranked Secondary Endpoint #7: Proportion of Participants With Mucosal Healing at Week 8 (Adalimumab 80/40 Versus Placebo).
Description: Mucosal healing defined as Endoscopy Subscore of 0 or 1 as assessed by flexible sigmoidoscopy. Possible scores range from 0-3 as follows:
  0 = Normal or inactive disease, 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 2 = Moderate disease (marked erythema, absent vascular pattern, friability, erosions), 3 = Severe disease (spontaneous bleeding, ulceration)
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 41.5 | 37.7
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80/40; Test type: Superiority or Other; p = 0.526, Chi-squared — [p-value comment as in outcome 2, analysis 1]

9. Secondary Outcome: Ranked Secondary Endpoint #8: Proportion of Participants With Rectal Bleeding Subscore Indicative of Mild Disease (<= 1) at Week 8 (Adalimumab 80/40 Versus Placebo).
Description: as for outcome 4
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 66.2 | 70.0
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80/40; Test type: Superiority or Other; p = 0.506, Chi-squared — [p-value comment as in outcome 2, analysis 1]

10. Secondary Outcome: Ranked Secondary Endpoint #9: Proportion of Participants With Physician's Global Assessment Subscore Indicative of Mild Disease (<= 1) at Week 8 (Adalimumab 80/40 Versus Placebo).
Description: as for outcome 5
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 46.9 | 53.8
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.264, Chi-squared — [p-value comment as in outcome 2, analysis 1]

11. Secondary Outcome: Ranked Secondary Endpoint #10: Proportion of Participants With Stool Frequency Subscore Indicative of Mild Disease (<= 1) at Week 8 (Adalimumab 80/40 Versus Placebo).
Description: as for outcome 6
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 37.7 | 36.2
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80/40; Test type: Superiority or Other; p = 0.797, Chi-squared — [p-value comment as in outcome 2, analysis 1]

12. Secondary Outcome: Ranked Secondary Endpoint #11: Proportion of IBDQ Responders at Week 8 (Adalimumab 160/80/40 Versus Placebo).
Description: Response per the Inflammatory Bowel Disease Questionnaire (IBDQ) defined as a >= 16-point increase from Baseline in total IBDQ score. The IBDQ is a 32-item questionnaire consisting of 4 dimensions: bowel-related symptoms, systemic function, social function, and emotional status. The responses to each question within each domain range from 1 (significant impairment) to 7 (no impairment), with total score ranging from 32 (very poor) to 224 (perfect health-related quality of life).
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 160/80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 57.7 | 60.8
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 160/80/40; Test type: Superiority or Other; p = 0.614, Chi-squared — [p-value comment as in outcome 2, analysis 1]

13. Secondary Outcome: Ranked Secondary Endpoint #12: Proportion of IBDQ Responders at Week 8 (Adalimumab 80/40 Versus Placebo).
Description: as for outcome 12
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Adalimumab 80/40
Number analyzed (Participants) | 130 | 130
Proportion of participants | 57.7 | 53.8
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80/40; Test type: Superiority or Other; p = 0.532, Chi-squared — [p-value comment as in outcome 2, analysis 1]

14. Secondary Outcome: Proportion of Participants With Clinical Remission Per Mayo Score at Week 52
Description: as for outcome 1
Time Frame: Week 52
Population: All randomized participants (enrolled under any version of the protocol) who received at least 1 dose of study drug were included in this intent-to-treat analysis. Nonresponder imputation (NRI) was used; participants who dose escalated to adalimumab 40 mg ew were considered nonresponders after their dose escalation.
Measure: Number; unit: Proportion of participants
Groups:
- Total: All subjects who received at least 1 dose of adalimumab or placebo
Arm/Group | Total
Number analyzed (Participants) | 575
Proportion of participants | 24.2

15. Secondary Outcome: Proportion of Participants With Clinical Remission Per Partial Mayo Score at Week 52
Description: Clinical remission per partial Mayo score is defined as a partial Mayo score <= 2 and no individual subscore > 1.
  The partial Mayo score is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 9 (severe disease) and is a composite of 3 subscores:
  Stool Frequency Subscore, Rectal Bleeding Subscore, and Physician's Global Assessment Subscore, each of which ranges from 0 (normal) to 3 (severe disease).
Time Frame: Week 52
Population: as for outcome 14
Measure: Number; unit: Proportion of participants
Arm/Group | Total
Number analyzed (Participants) | 575
Proportion of participants | 28.3

16. Secondary Outcome: Proportion of Participants With Clinical Response Per Mayo Score at Week 52
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 14
Measure: Number; unit: Proportion of participants
Arm/Group | Total
Number analyzed (Participants) | 575
Proportion of participants | 42.6

17. Secondary Outcome: Proportion of Participants With Clinical Response Per Partial Mayo Score at Week 52
Description: Clinical response per partial Mayo score is defined as a decrease in partial Mayo score of >= 2 points and >= 30% from Baseline, plus either a decrease in rectal bleeding subscore of >= 1 point or an absolute rectal bleeding subscore of 0 or 1.
  The partial Mayo Score is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 9 (severe disease) and is a composite of 3 subscores:
  Stool Frequency Subscore, Rectal Bleeding Subscore, and Physician's Global Assessment Subscore, each of which ranges from 0 (normal) to 3 (severe disease).
Time Frame: Week 52
Population: All randomized participants (enrolled under any version of the protocol) who received at least 1 dose of study drug were included in this intent-to-treat analysis. Nonresponder imputation (NRI) was used; subjects who dose escalated to adalimumab 40 mg ew were considered nonresponders after their dose escalation.
Measure: Number; unit: Proportion of participants
Arm/Group | Total
Number analyzed (Participants) | 575
Proportion of participants | 41.6

18. Secondary Outcome: Proportion of Participants With Mucosal Healing at Week 52
Description: as for outcome 3
Time Frame: Week 52
Population: as for outcome 14
Measure: Number; unit: Proportion of participants
Arm/Group | Total
Number analyzed (Participants) | 575
Proportion of participants | 36.5

19. Secondary Outcome: Proportion of Participants With Rectal Bleeding Subscore Indicative of Mild Disease (<= 1) at Week 52
Description: as for outcome 4
Time Frame: Week 52
Population: as for outcome 14
Measure: Number; unit: Proportion of participants
Arm/Group | Total
Number analyzed (Participants) | 575
Proportion of participants | 47.0

20. Secondary Outcome: Proportion of Participants With Physician's Global Assessment Subscore Indicative of Mild Disease (<= 1) at Week 52
Description: as for outcome 5
Time Frame: Week 52
Population: as for outcome 14
Measure: Number; unit: Proportion of participants
Arm/Group | Total
Number analyzed (Participants) | 575
Proportion of participants | 41.7

21. Secondary Outcome: Proportion of Participants With Stool Frequency Subscore Indicative of Mild Disease (<= 1) at Week 52
Description: as for outcome 6
Time Frame: Week 52
Population: as for outcome 14
Measure: Number; unit: Proportion of participants
Arm/Group | Total
Number analyzed (Participants) | 575
Proportion of participants | 36.5

22. Secondary Outcome: Proportion of Participants With Clinical Remission Per Mayo Score at Week 52 Among Participants Who Were Systemic Corticosteroid-free at Week 52
Description: as for outcome 1
Time Frame: Week 52
Population: All randomized participants enrolled under any version of the protocol who took systemic corticosteroids (CS) at Baseline, received at least 1 dose of study drug, and were systemic CS-free at Week 52 were included. Nonresponder imputation was used; participants who dose escalated to adalimumab 40 mg ew were considered nonresponders post-escalation.
Measure: Number; unit: Proportion of participants
Arm/Group | Total
Number analyzed (Participants) | 316
Proportion of participants | 41.5

ADVERSE EVENTS:
Time Frame: Adverse event data are presented through Week 8 for the placebo, adalimumab 80/40, and adalimumab 160/80/40 groups. Adverse event data are presented through Week 52 for the Any Adalimumab group.
Description: Adverse events reported in the "Any Adalimumab" group include those reported in the "Adalimumab 80/40" and "Adalimumab 160/80/40" groups (during the double-blind phase) plus adverse events reported during open-label adalimumab treatment.
Groups:
- Placebo: Treatment group received placebo at Weeks 0, 2, 4, and 6. Adverse events include those reported prior to dosing at Week 8.
- Adalimumab 80/40: Treatment group received 80 mg at Week 0, 40 mg at Week 2, and 40 mg every other week starting at Week 4. Adverse events include those reported prior to dosing at Week 8.
- Adalimumab 160/80/40: Treatment group received 160 mg at Week 0, 80 mg at Week 2, and 40 mg every other week starting at Week 4. Adverse events include those reported prior to dosing at Week 8.
- Any Adalimumab: Treatment group received at least 1 dose of adalimumab during the study. Adverse events include those reported from the first dose of adalimumab during the double-blind or open-label period.
Arm/Group | Placebo | Adalimumab 80/40 | Adalimumab 160/80/40 | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 17/223 | 5/130 | 9/223 | 76/557
Other Adverse Events (participants affected / at risk) | 34/223 | 30/130 | 34/223 | 210/557
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=223) | Adalimumab 80/40 (N=130) | Adalimumab 160/80/40 (N=223) | Any Adalimumab (N=557)
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 13 | 3 | 4 | 34 — As this was a study in subjects with ulcerative colitis as the underlying disease, the event term of "colitis ulcerative" refers to worsening of the disease (i.e., flare).
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Abscess rupture (Infections and infestations) | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 2
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Personality disorder (Psychiatric disorders) | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 2
Nasal septal operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 3
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=223) | Adalimumab 80/40 (N=130) | Adalimumab 160/80/40 (N=223) | Any Adalimumab (N=557)
Colitis ulcerative (Gastrointestinal disorders) | 8 | 7 | 9 | 85 — As this was a study in subjects with ulcerative colitis as the underlying disease, the event term of "colitis ulcerative" refers to worsening of the disease (i.e., flare).
Headache (Nervous system disorders) | 16 | 9 | 7 | 47
Nausea (Gastrointestinal disorders) | 4 | 4 | 4 | 31
Fatigue (General disorders) | 5 | 2 | 9 | 33
Nasopharyngitis (Infections and infestations) | 4 | 6 | 6 | 53
Upper respiratory tract infection (Infections and infestations) | 6 | 6 | 3 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.